CLINICAL TRIAL: NCT04807270
Title: Efficacy of Two Different Platelet Rich Plasma Methods in Patients With Knee Osteoarthritis: A Randomized Controlled Study
Brief Title: PRP Effectiveness in Knee Osteoarthritis
Acronym: PRP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Sinan GOK, MD, Sub-Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Istanbul Universty PRP
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; platelet rich plasma
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T-LAB / PRP KIT (Active Comparator): In the first group, Platelet-rich plasma (PRP) prepared with T-LAB / PRP KIT injection in 3 sessions will be applied.
  Interventions: Other: Intra-articular T-LAB / PRP KIT injection
- T-LAB / PRP INJECTION SYRINGE (Active Comparator): In the first group, Platelet-rich plasma (PRP) prepared with T-LAB / PRP INJECTION SYRINGE injection in 3 sessions will be applied.
  Interventions: Other: Intra-articular T-LAB / PRP INJECTION SYRINGE injection
- SALINE (Active Comparator): In the first group, Platelet-rich plasma (PRP) prepared with SALINE injection in 3 sessions will be applied.
  Interventions: Other: Intra-articular SALINE injection

INTERVENTIONS:
Other: Intra-articular T-LAB / PRP KIT injection — Intra-articular 3 ml T-LAB / PRP KIT injection in 3 sessions will be applied. As a home exercise program, hamstring and quadriceps stretching, quadriceps isometric strengthening, short arc terminal extension exercises will be given at least three days a week with 3 sets of 10 repetitions.
  Arms: T-LAB / PRP KIT
Other: Intra-articular T-LAB / PRP INJECTION SYRINGE injection — Intra-articular 3 ml T-LAB / PRP INJECTION SYRINGE injection in 3 sessions will be applied. As a home exercise program, hamstring and quadriceps stretching, quadriceps isometric strengthening, short arc terminal extension exercises will be given at least three days a week with 3 sets of 10 repetitions.
  Arms: T-LAB / PRP INJECTION SYRINGE
Other: Intra-articular SALINE injection — Intra-articular 3 ml SALINE injection in 3 sessions will be applied. As a home exercise program, hamstring and quadriceps stretching, quadriceps isometric strengthening, short arc terminal extension exercises will be given at least three days a week with 3 sets of 10 repetitions.
  Arms: SALINE

SUMMARY:
The aim of our study is to determine the effects of intra-articular Platelet Rich Plasma (PRP) prepared with two different techniques on pain intensity, functional status, quality of life, functional balance and femoral cartilage thickness in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common form of chronic joint disease. Platelet Rich Plasma (PRP) is an injection therapy used to treat chronic painful musculoskeletal conditions, including knee OA. In this prospective, randomized controlled, single blind, interventional study, a total of 75 patients with stage 2-3 knee osteoarthritis according to the kellgren lawrence classification who meet the eligibility criteria will be enrolled in the study. Eligible participants will be randomly assigned to one of the three groups using computer-generated random numbers.The patients to be included in the study will be randomized into three groups and the first group will be given platelet-rich plasma (PRP) prepared with T-LAB / PRP KIT, the second group will be given PRP prepared with T-LAB PRP INJECTION SYRINGA, and the third group will be given saline injection. Home exercise program for knee osteoarthritis will be given to all three groups and the exercise program will be followed by weekly phone calls. During the follow-up period, patients will be asked to continue their current medical treatments, not to make changes in their activities of daily living. Participants are going to evaluate before injection, and at the 1-month follow-up and 6-month follow-up using the visual analog scale (VAS) scores for pain during activity, at rest, and at night, with the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) change in pain, stiffness and physical function score, the change in the Timed Up and Go Test (TUG) time, change in femoral cartilage thickness measurement by ultrasound and the change in the patient's daily activities with the numerical global patient assessment scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic symptomatic knee pain between the ages of 30-75 years
* Presence of Kellgren-Lawrence stage 2-3 osteoarthritis on current anterior-posterior knee radiographs
* Functional ambulation scale stage 4-5

Exclusion Criteria:

* Intra-articular knee injection within the last six months
* History of severe trauma to the knee within the past six months
* Concomitant severe meniscus or ligament injury, surgery applied to the knee area
* Presence of severe effusion, inflammatory joint disease, infection, hematological and oncological disease in the knee.
* Having a bleeding disorder and / or using warfarin
* Kellgren-Lawrence stage 1 or stage 4 osteoarthritis on current anterior-posterior knee radiographs
* Presence of cardiac or systemic disease that may affect exercise
* The presence of neurological disease and psychiatric disease such as Parkinson's disease, stroke history that may affect balance
* Body Mass Index ≥35 kg / m²

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-03-22 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline activity pain score at 1-months and 6-months | Baseline, 1-month, 6-month
  Visual Analogue Scale-Activity pain (0-10 point). Higher scores mean a worse outcome

SECONDARY OUTCOMES:
Change from baseline rest pain score at 1-months and 6-months | Baseline, 1-month, 6-month
  Visual Analogue Scale-Rest pain (0-10 point). Higher scores mean a worse outcome
Change from baseline night pain score at 1-months and 6-months | Baseline, 1-month, 6-month
  Visual Analogue Scale-Night pain (0-10 point). Higher scores mean a worse outcome
Change from baseline pain, stiffness and physical function at 1-months and 6-months | Baseline, 1-month, 6-month
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) measures knee pain, stiffness, and physical function. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The sum of the scores for the three subscales gives a total WOMAC score. High scores are associated with more pain, stiffness, and poor function, while low scores indicate well-being.
Change from baseline functional balance at 1-months and 6-months | Baseline, 1-month, 6-month
  The Timed Up and Go test requires the person to stand up from a standard chair in which they are sitting, walk 3 m at a comfortable speed to the marked place on the floor, turn around, walk backwards to the starting point and return to the sitting position in the chair. The time taken for the person to complete the test is measured in seconds. The timing of the test is related to the function.
Change from baseline femoral cartilage thickness measurement by ultrasound at 6 months | Baseline, 6-month
  Distal femoral cartilage thickness will be evaluated by the same clinician using the MyLab60 model ultrasonography device and high-resolution 7-12 MHz linear probe available in our clinic. During the measurement, patients will be positioned in the prone position with their knees in full flexion and ankles in neutral to examine the distal femoral cartilage, and the probe will be placed in the axial position in the suprapatellar area at the outer edge of the patella. After the distal femoral cartilage is anechogenically imaged between the hyperechogenic bony cortex and suprapatellar fat, the distance between the thin hyperechoic line of the synovial cavity on the stratified face and the hyperechoic sharp line on the bony face of the cartilage will be measured and recorded as the thickness of the cartilage. Cartilage thickness measurements for each intervention knee will be recorded by recording three measurements from the midpoint: lateral condyle, intercondylar area and medial condyle.

CONTACTS AND LOCATIONS:
Overall Officials: Demirhan Diracoglu, Prof., Study Director — Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation; Ekin I Sen, Asst. Prof., Principal Investigator — Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Fatıh, Turkey (Türkiye)